CLINICAL TRIAL: NCT03730597
Title: Influenze of Glenosphere Size in Scapular Notch Development. Randomized Study Comparing 42 to 38 ECC
Brief Title: Glenosphere Size and Scapular Notch in RSA, Prospective Randomized Study
Acronym: GSSNRSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital del Mar (Other)
Responsible Party: Principal Investigator, Carlos Torrens, Head of Shoulder Unit, Hospital del Mar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Torrens.00; CTorrens (Other: HMar)
Record Dates: First submitted 2018-10-31; First posted 2018-11-05 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2018-10

CONDITIONS: Total Shoulder Arthroplasty

STUDY DESIGN:
Intervention Model Description: randomized study
Who Masked: Outcomes Assessor
Masking Description: blinded to purpose of study and to randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- glenosphere 42 (Active Comparator): patients receiving a reverse shoulder arthroplasty with a glenosphere sized 42. reverse shoulder prosthesis implantation X-Ray analysis to detect scapular notch
  Interventions: Device: reverse shoulder arthroplasty
- glenosphere 38 ECC (Active Comparator): patients receiving a reverse shoulder arthroplasty with a glenosphere sized 38 ECC reverse shoulder prosthesis implantation X-Ray analysis to detect scapular notch
  Interventions: Device: reverse shoulder arthroplasty

INTERVENTIONS:
Device: reverse shoulder arthroplasty — prosthesis implantation
  Other Names: Delta X-tend

SUMMARY:
Scapular notch can be reduced by using bigger glenospheres but in some patients it cannot be implanted because of small size. If small size of glenosphere is used then scapular notch may increase. To improve that situation, eccentricity has been added to some glenospheres to increase glenoid overhanging. The objective is to assess if eccentricity can avoid scapular notch as effectively as bigger glenospheres.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing reverse shoulder prosthesis because of rotator cuff disordes andacute fractures

Exclusion Criteria:

* patients with previous surgery
* patients with deltoid deficiency
* patients with acute infection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2016-09-09 (Actual); Study Completion 2016-09-09 (Actual)

PRIMARY OUTCOMES:
scapular notch development | two years
  X-ray assessment of scapular notch development

IPD SHARING:
Plan to Share IPD: No